CLINICAL TRIAL: NCT05018156
Title: Pilot Implementation Study of a Default Genetics Referral Process for Patients With Young-Onset Colorectal Cancer
Brief Title: Default Genetics Referrals for Young-Onset Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Kelsey Lau-Min, MD, Hematology/Oncology Fellow, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 849320
Record Dates: First submitted 2021-08-06; First posted 2021-08-24 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Default Genetics Referral Process (Experimental)
  Interventions: Behavioral: Default Genetics Referral Process

INTERVENTIONS:
Behavioral: Default Genetics Referral Process — Patients and their oncology providers will be notified of their eligibility for a cancer genetics referral, with an option to opt out if they are not interested in proceeding. Everyone else will be automatically referred to their local hospital's cancer genetics program for contact and scheduling. Standard genetic counseling, testing, and results disclosure will take place, including usual methods of payment and insurance coverage for testing.

SUMMARY:
The investigators will perform a pilot implementation study of a default genetics referral process among patients with young-onset CRC diagnosed between ages 40 and 49.

DETAILED DESCRIPTION:
The incidence of young-onset colorectal cancer (CRC) - defined as a diagnosis of CRC prior to age 50 - has increased at alarming rates in recent years. Over 75% of cases occur in patients diagnosed between 40-49 years old, a group that is not traditionally included in young adult cancer initiatives tailored only to patients up to 39 years of age. Young age of CRC onset is a defining feature of hereditary CRC syndromes; as such, the National Comprehensive Cancer Network and American College of Medical Genetics and Genomics recommend germline genetics evaluations for all patients diagnosed with CRC under the age of 50. However, multiple studies have shown suboptimal rates and racial and socioeconomic disparities in guideline-recommended genetics evaluations.

In this pilot implementation study, the investigators aim to develop, implement, and evaluate the effects of a default genetics referral process among patients with young-onset CRC diagnosed between 40-49 years old. The investigators hypothesize that by applying defaults, or pre-selected choices, to minimize the cognitive effort that patients and clinicians use to make decisions, default referrals will improve rates of genetics referrals while reducing existing racial and socioeconomic disparities. The investigators will implement this intervention at five academic and community hospitals within Penn Medicine that serve a racially, socioeconomically, and geographically diverse patient population. The investigators will use an automated electronic health record-based algorithm to identify eligible patients, after which default referrals for genetic risk evaluation will be made unless patients or their oncology clinicians opt out. The investigators will rigorously evaluate the impact of this default genetics referral process using mixed methods leveraging models and frameworks from the field of implementation science.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with colon or rectal adenocarcinoma
* Between 40-49 years old at the time of index cancer diagnosis
* At least two visits at Penn Medicine for the evaluation or treatment of the index cancer

Exclusion Criteria:

* Diagnosis of in situ cancer
* Known genetic predisposition to cancer
* Genetic testing after index cancer diagnosis

Ages: 40 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Genetics referrals | 3 months
  The number of patients who are ultimately referred to genetics divided by the total number of eligible patients

SECONDARY OUTCOMES:
Scheduled genetics evaluations | 3 months
  The proportion of genetics evaluations that are scheduled divided by the total number of genetics referrals
Completed genetics evaluations | 3 months
  The proportion of genetics evaluations that are completed divided by the total number of scheduled genetics evaluations
Genetic testing | 3 months
  The proportion of genetics evaluations that result in genetic testing divided by the total number of completed genetics evaluations

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No